CLINICAL TRIAL: NCT07168694
Title: Retrospective, Multicenter, Non-interventional (Observational) Study With the Aim to Describe the Impact of Siponimod Treatment in a Real-world SPMS Population in Russia
Brief Title: A Real-world Study About the Impact of Siponimod Treatment on Secondary Progressive Multiple Sclerosis Patients in Russia
Acronym: EMBOSSES
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312ARU02
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Siponimod; Treatment of multiple sclerosis; Real-world clinical data
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Siponimod Cohort: Adult patients with SPMS who were treated with siponimod.

SUMMARY:
The main aim of the study was to describe the demographic and clinical characteristics of patients with secondary progressive multiple sclerosis (SPMS) who were receiving siponimod therapy in Russia. This study analyzed data from outpatient records/medical records collected across 11 Russian multiple sclerosis (MS) centers. Data collection was carried out from April 16, 2024 to September 26, 2024.

ELIGIBILITY:
Inclusion criteria:

* Documented diagnosis of SPMS, with or without relapses.
* Treatment with siponimod for at least 6 months.

Exclusion criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Demographics: Number of Patients by Age | Baseline
Demographics: Number of Patients by Gender | Baseline
Time Between MS Diagnosis and Treatment Initiation | Baseline
Time Between SPMS Diagnosis and Treatment Initiation | Baseline
Time Between First Symptoms and Treatment Initiation | Baseline
Number of Patients by Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * MS symptoms
  * Magnetic resonance imaging (MRI) performed (yes/no)
  * Number of contrast-enhancing lesions on T1-weighted images (WI) (Gd+T1 lesions): absent, single, or multiple lesions
  * CYP2C9 isoenzyme genotype
Number of Patients Categorized by Type of Treatment Received Before Initiation of Siponimod | Baseline
  Treatment categories included glucocorticosteroids, cytostatics, and disease-modifying treatments (DMTs).
Number of Patients by DMT Received Before Initiation of Siponimod | Baseline
Duration of the Washout Period After Other DMTs and Before Initiation of Siponimod | Baseline
Number of Patients by Reason for Switching From Other DMTs to Siponimod | Baseline
Duration of Siponimod Therapy | Up to 2 years

SECONDARY OUTCOMES:
Change From Baseline in Expanded Disability Status Scale (EDSS) Score | Baseline and Months 6, 12, 18, 24
  The EDSS is a tool used by doctors to measure disability in MS patients and monitor changes in the level of disability over time. It focuses on rating 7 functional systems: visual function, brainstem symptoms (speech, swallowing, rapid eye movement), pyramidal (muscle strength and movement), cerebellar (coordination and balance), sensory, bowel and bladder function, and higher cerebral functions (thinking and memory). These ratings are then used in conjunction with observations and information concerning gait and use of assistive devices to rate the EDSS. EDSS scores range from 0 (normal) up to 10 (death due to MS).
Percentage of Patients With Confirmed Disability Progression Over 6 Months (6m-CDP) Based on the EDSS Score | Months 6, 12, 18, 24
  Confirmed disability progression is determined when a patient shows a sustained or increased EDSS score compared to the date of the first documented worsening of neurological function, assessed at least 6 months later, provided there are no relapses during the assessment period. A clinically meaningful worsening of neurological function is defined as an increase in EDSS score of 1.5 points for patients with a baseline EDSS of 0, 1.0 point for those with a baseline EDSS of 1.0 to 5.5, or 0.5 points for patients with a baseline EDSS of 6.0.
Number of Patients With MS Relapses | Baseline
Annualized Relapse Rate (ARR) | 1 and 2 years before siponimod initiation and 6, 12, 18, and 24 months after siponimod treatment
Change in ARR From 1 Year Before Siponimod Initiation to 6, 12, 18, and 24 Months After Siponimod Treatment | 1 year before siponimod initiation and 6, 12, 18, and 24 months after siponimod treatment
Number of Patients With MRI Signs of MS After Siponimod Treatment | Months 6, 12, 18, 24
  MRI signs included:
  * Contrast-enhancing lesions on T1-WI (Gd+T1 lesions): absent, single, or multiple lesions
  * New/enlarged lesions on T2-WI or contrast-enhancing lesions on T1-WI (Gd+T1 lesions)
Number of Patients by Reason for Stopping Siponimod Treatment | Months 6, 12, 18, 24
Number of Patients With Siponimod-related Adverse Events | Months 6, 12, 18, through study follow-up, up to approximately 24 months
Number of Patients With Siponimod-related Serious Adverse Events | Months 6, 12, 18, through study follow-up, up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States